CLINICAL TRIAL: NCT04387214
Title: The Impact of COVID-19 Pandemic on the Academic Performance of Veterinary Medical Students and Researchers
Brief Title: COVID-19 Pandemic and Academic Performance of Veterinary Students
Status: Completed | Type: Observational
Sponsor: South Valley University (Other)
Responsible Party: Principal Investigator, Mohamed Mahdy, Principal Investigator, South Valley University
Other Study IDs: 1-2020
Record Dates: First submitted 2020-05-12; First posted 2020-05-13 (Actual); Last update posted 2020-09-09 (Actual); Status verified 2020-09

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Veterinary students and researchers
  Interventions: Other: survey

INTERVENTIONS:
Other: survey — online survey

SUMMARY:
The study aims to analyze the effect of COVID-19 pandemic on the academic performance of veterinary students, veterinarians, and researchers during the lockdown.

ELIGIBILITY:
Inclusion Criteria:

* Veterinary students and researchers

Exclusion Criteria:

-

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Veterinary students and researchers
Sampling Method: Probability Sample
Enrollment: 1426 (Actual)
Dates: Start 2020-04-13 (Actual); Primary Completion 2020-08-10 (Actual); Study Completion 2020-08-10 (Actual)

PRIMARY OUTCOMES:
Measure the effect of COVID-19 pandemic on the academic performance of veterinary medical students | 13/4/2020 - 10/8/2020
  An online questionnaire (Question:How did COVID-19 pandemic affect your study/ research?. Response: Greatly affected, Moderately affected, slightly affected, Not affected
Measure the average studying time | 13/4/2020 - 10/8/2020
  Open question: How many hours do you spend in on-line learning?
Evaluate on-line education during COVID-19 pandemic lockdown | 13/4/2020 - 10/8/2020
  Question:How do you rate on-line education? Answer on 1-10 scale, 1 is the lowest evaluation and 10 is the highest evaluation
Evaluate on-line education in practical lessons during COVID-19 pandemic lockdown | 13/4/2020 - 10/8/2020
  Question:How do you rate on-line education in practical lessons? Answer on 1-10 scale, 1 is the lowest evaluation and 10 is the highest evaluation

CONTACTS AND LOCATIONS:
Locations (1):
- South Valley University, Qina, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Published paper — https://www.frontiersin.org/articles/10.3389/fvets.2020.594261/abstract